CLINICAL TRIAL: NCT04828291
Title: Optimizing Daily Mindfulness Interventions Using Peer Support to Increase Well-Being in First-Year Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pitzer College (Other)
Responsible Party: Principal Investigator, Marcus Rodriguez, Co-PI, Pitzer College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3661
Record Dates: First submitted 2021-03-12; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: OMI, OMI+, Control Group
MeSH Terms: conditions — Parkinson Disease 13

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online Mindfulness Intervention (OMI) (Experimental): Before beginning the daily practices, this group will be introduced to the OMI via an online platform and answer any questions about the practice. Then, each day, this group will be guided through a series of mindfulness practices offered online (www.bemindfulonline.com) delivered on their smartphones or laptops.
  Interventions: Behavioral: Benign Behavioral Interventions
- OMI paired with peer support (OMI+) (Experimental): Before beginning the daily OMI, in addition to being briefed, this group will be paired with a peer to be in touch with and guide and support each other in this process. Then they will start the OMI program and will follow parallel instructions as the OMI group. The peer support will include five brief (30-minute) weekly meetings to support and encourage each other to continue practicing mindfulness and to complete the online intervention. Each week we will provide prompts and topics for participants to discuss and at the end of each meeting, participants will then complete a short, 5-10 minute post-meeting survey to assess the well-being and attitudes of their partner (see additional materials for meeting prompts and post-meeting survey questions). The first of these meetings will occur on Day 8, and subsequent weekly meetings during the intervention period will be scheduled based on the shared availability of both participants in each pair.
  Interventions: Behavioral: Benign Behavioral Interventions
- Active control receiving cognitive exercises (Active Comparator): Instead of the OMI, this group will be receiving cognitive exercises in the intervention period.
  Interventions: Behavioral: Benign Behavioral Interventions

INTERVENTIONS:
Behavioral: Benign Behavioral Interventions — This project will use a Randomized Control Trial (RCT) design and Daily Reconstruction Method (DRM8) to model the effects of the OMI on dynamic changes in first-year undergraduate and graduate students' well-being over time. The intervention will take place over the course of 46 days, with a 7- day follow up assessment taking place one month after the intervention. People will complete surveys through an online link leading to Qualtrics.com.

SUMMARY:
This project aims to examine the effect of a self-guided, evidence-based, online mindfulness intervention on well-being among first-year undergraduates at the 5 Claremont Colleges (5C's) and graduate students in the community. Additionally, it explores the feasibility and efficacy of peer support (pairs) as an adjunctive treatment component to enhance engagement and treatment effects, including social-connectedness, well- being, academic outcomes, and anxiety. Findings will provide insight into effective ways to (1) support students at The Claremont Colleges, and (2) leverage technology and peer support to implement mental health initiatives that are cost-effective, easily transportable, and scalable in low-resource settings.

ELIGIBILITY:
Inclusion Criteria:

* all participants must be either a first-year undergraduate student or a graduate student. Participants must be 18 years or older.

Exclusion Criteria:

* all participants must be either a first-year undergraduate student or a graduate student. Participants must be 18 years or older.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Five Facet Mindfulness Questionnaire (FFMQ) | Baseline to Day 46
  The FFMQ is a self-reported, instrument assessing mindfulness based on five factors that represent elements of mindfulness ( observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience). Possible scores range from 1 (never or very rarely true) to 5 (very often or always true).
  Reference: Bohlmeijer, E., P. M. ten Klooster, et al. (2011). "Psychometric properties of the five facet mindfulness questionnaire in depressed adults and development of a short form." Assessment 18(3): 308-320

SECONDARY OUTCOMES:
Sample Attrition | Baseline to Day 46
  Completion rate or drop out rate comparing OMI group versus OMI+ group in a 46 day longitudinal study.
PERMA (Overall Well Being) | Day 0-46
  The self-reported measure consists of 23 items. The health, negative emotion, loneliness, and overall happiness questions act as filler questions and provide more information; for briefness, the 15 PERMA questions (3 per PERMA domain) could be used, but we recommend using the full measure.
  Reference: Butler, J., & Kern, M. L. (2016). The PERMA-Profiler: A brief multidimensional measure of flourishing. International Journal of Wellbeing, 6(3), 1-48. doi:10.5502/ijw.v6i3.1

OTHER OUTCOMES:
Self-Report Health (SF-36) | Baseline
  SF-36 is a self-reported instrument assessing easily administered quality-of-life measures which consists of 8 subscales. These measures rely upon patient self-reporting and are now widely utilized by managed care organizations and by Medicare for routine monitoring and assessment of care outcomes in adult patients.
  Reference: Ware, IE. Jr., Snow, K.K, Kosinski, M., & Gandek, B. (1993). SF-36 Health Survey. Manual and Interpretation Guide. Boston, MA: Nimrod Press.
Academic Motivation Scale | Day 38
  The Academic Motivation Scale (AMS) is a validated, self-reported, seven point Likert type item scale that measures Intrinsic, extrinsic, and Amotivation in education. Possible scores range from 1 (does not correspond at all) to 7 (corresponds exactly).
  Reference: Vallerand, R. J., Pelletier, L. G., Blais, M. R., Brière, N. M., Senécal, C. B., & Vallières, É. F. (1993). Academic motivation scale (ams-c 28) college (cegep) version. Educ Psychol Meas, 52, 1003-17.

CONTACTS AND LOCATIONS:
Locations (1):
- Claremont Graduate University, Claremont, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR